CLINICAL TRIAL: NCT07386444
Title: Effects of Inspiratory Muscle Training Among Breast Cancer Patients Undergoing Active Treatment (IMACT)
Brief Title: Inspiratory Muscle Training for Breast Cancer Patients on Chemotherapy
Acronym: IMACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Dharini Bhammar, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OSU-25238; NCI-2026-00179 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Early Stage Breast Carcinoma; Dyspnea
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blinded to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (low-intensity IMT) (Active Comparator): Patients complete three sets of fifteen repetitions per session of low-intensity IMT over 15-20 minutes four days a week for 8 weeks.
  Interventions: Behavioral: Inspiratory muscle training
- Arm 2 (high-intensity IMT) (Experimental): Patients complete three sets of fifteen repetitions per session of high-intensity IMT over 15-20 minutes four days a week for 8 weeks.
  Interventions: Behavioral: Inspiratory muscle training

INTERVENTIONS:
Behavioral: Inspiratory muscle training — Training of respiratory muscles

SUMMARY:
This clinical trial studies whether breathing exercises for the muscles that help with breathing air in, inspiratory muscle training (IMT), works to improve breathing muscle strength, shortness of breath, and physical activity levels in women who are receiving chemotherapy for early-stage breast cancer (BC). Cancer and/or treatments for BC can directly result in muscle wasting that involves breathing muscles, skeletal muscles or heart muscles. Pain, weakness, shortness of breath, and side effects of cancer treatment may lead to lower physical activity levels. IMT involves breathing exercises using a small hand-held device. The device makes it a little harder to breathe in, which may help strengthen breathing muscles. IMT may be an effective way to improve breathing muscle strength, shortness of breath, and physical activity levels in women who are receiving chemotherapy for early-stage BC.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE: To investigate the effects of 8 weeks of IMT on inspiratory muscle strength, exertional dyspnea, and physical activity levels among women undergoing chemotherapy for BC.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients complete three sets of fifteen repetitions per session of low-intensity IMT over 15-20 minutes four days a week for 8 weeks.

ARM 2: Patients complete three sets of fifteen repetitions per session of high-intensity IMT over 15-20 minutes four days a week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Within 3 weeks of starting chemotherapy for an early-stage breast cancer diagnosis
* Able to exercise independently without needing support
* Ability to read, speak, understand English

Exclusion Criteria:

* Metastatic breast cancer
* Unwilling or unable to follow protocol requirements
* Any significant health condition which in the investigator's opinion increases the risks of participation or makes the participant unsuitable for the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2026-02-19 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum inspiratory pressure | Baseline to 8 weeks
  Measure of the strength of the inspiratory muscles. Units: cm H20

SECONDARY OUTCOMES:
Physical activity levels | Baseline to 8 weeks
  Number of steps/day averaged weekly.
Modified Medical Research Council Dyspnea scale rating | Baseline to 8 weeks
  Patients will indicate the extent to which their dyspnea affects mobility using a one question 1-5 scale; higher scores indicate greater respiratory disability.
Dyspnea 12 score | Baseline to 8 weeks
  Questionnaire consists of 12 descriptor items such as "I feel short of breath" and "my breathing is uncomfortable" with each item rated on a scale of none (0), mild (1), moderate (2), or severe (3). Individual items are summed to generate a total score (0 to 36), with a higher score indicating worse dyspnea
RAND-36 Quality of life | Baseline to 8 weeks
  8 subdomains will be scored 0-100 with higher scores reflecting better perceived quality of life.
FACIT-F | Baseline to 8 weeks
  Version 4 is a 40-item measure that will be used to assess self-reported fatigue and its impact on daily activities and function over the past 7 days. It is a 5-point Likert-type scale with five subdomains including physical well-being, social/family well-being, emotional well-being, functional well-being, and fatigue yielding a total score from 0-52.

OTHER OUTCOMES:
Relative dose intensity of chemotherapy | At 8 weeks
  Will record the relative dose intensity of chemotherapy for each participant. The relative dose intensity will be averaged for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Dharini M Bhammar, MBBS, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make deidentified data freely available if requested. The privacy and rights of the participants will be protected.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available after data collection is complete for up to 3 years.
Access Criteria: Deidentified data will be made available on request following approved data use agreements between institutions.

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu